CLINICAL TRIAL: NCT02731495
Title: Effect of Green Tea Epigallocatechin -3-gallate Supplementation on Traumatic Brain Injury Patients' Outcomes
Brief Title: Effect of Epigallocatechin -3-gallate Supplementation in Traumatic Brain Injury Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Collaborators: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Associate professor, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24513540293
Record Dates: First submitted 2016-02-17; First posted 2016-04-07 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EGCG (Experimental): Participants were randomly divided based on age, sex and severity of TBI in two groups. Randomization lists was computer-generated by a statistician and participants, project managers and employees at the clinic are completely unaware (blind) about intervention and control groups. At the first visit, baseline data were gathered and patients received EGCG supplement was in the form of 400 mg oral capsules with a purity of 80% catechin. EGCG powder of each capsule was dissolved in 10 ml deionized water and given to patients via gavage (1 capsule per day) for a week.
  Interventions: Dietary Supplement: EGCG
- Placebo (Placebo Comparator): Placebo group only received 10 ml of deionized water via gavage for a week.
  Interventions: Dietary Supplement: Placebo (deionized water)

INTERVENTIONS:
Dietary Supplement: EGCG — EGCG (Epigallocatechin -3-gallate)
  Arms: EGCG
Dietary Supplement: Placebo (deionized water)
  Arms: Placebo

SUMMARY:
Traumatic brain injury is the leading cause of death and disability in young adults. Green tea Epigallocatechin -3-gallate (EGCG) supplementation might favorably influenced many of the processes mention in the secondary insult of TBI including neuroinflammation and antioxidative damages.

The investigators aim to investigate whether treatment with Epigallocatechin -3-gallate favorably affect outcomes in traumatic brain injury patients. Therefore, in the current randomized double-blind clinical trial, 30 patients (15 patients in each group) with moderate to severe head trauma admitted to university hospital intensive care unit will included. Patients will either receive a daily oral dose of 400 mg EGCG or placebo for 7 days. The major outcomes includes duration of mechanical ventilation, Glasgow Coma Scale (GCS), and S100 protein level.

DETAILED DESCRIPTION:
Male patients (16-65 year old) who admitted to a university hospital intensive care unit with moderate to severe Traumatic Brain Injury (TBI) were enrolled using consecutive sampling. Inclusion criteria were GCS of 4-12, enteral nutrition started in 24 hours after admission, having mechanical ventilation. The procedure and protocol of the study was approved by the Ethic Committee of Tehran University of Medical Sciences. Written informed consent were obtained from patient's relative. After recording anamnesis, patients were examined physically. Urgent actions were done, simple radiography were taken from skull and CT-scan were performed if it is necessary. Patients who had internal bleeding, obvious fractures in their limbs, history of metabolic or psychiatric disorder, alcohol or drug dependency, underlying diseases, or vegetarian diet would be excluded from the study. Patients' base line information including age, sex, vital signs, GCS, clinical symptoms at time of reception, diagnosis based on CT-scan, type of treatment (medicinal or surgical) and surgical area of body were recorded. patients were then divided into two experimental groups: (1) receiving epigallocatechin gallate (EGCG) supplement (case group, n = 15) and (2) receiving placebo (control group, n = 15). EGCG supplement was in the form of 400 mg oral capsules with a purity of 80% catechin. EGCG powder of each capsule was dissolved in 10 ml deionized water and given to patients via gavage (1 capsule per day) for a week. Placebo group only received 10 ml of deionized water via gavage for a week. During that week, GCS of patients was recorded by a neurosurgery resident who was blinded. For seven days, vital signs, glucose, hematocrit, haemoglobin, platelet were recorded every day at 9:00 a.m. Duration of the connection to mechanical ventilation was also recorded.

In order to analyze serum S100B protein level, 5 ml serum was taken from patients at 1st day and 8th day of the admission and stored at -80⁰C. Human S100B ELISA kit was used to quantify the level of S100B protein.

Statistical analysis

distribution of all continuous variables was assessed using Kolmogorov-Smirnov test. Normal distributed variables were compared by independent samples t-test. Not-normal distributed variables were assessed by Wilcoxon-Mann-Whitney U-test. P value less than .05 would be considered as statistically significant for all tests. Data were analyzed using SPSS Statistics version 21 (SPSS Inc., Chicago, USA).

ELIGIBILITY:
Inclusion Criteria:

* GCS of 4-12
* enteral nutrition started in 24 hours after admission
* having mechanical ventilation.

Exclusion Criteria:

* internal bleeding
* obvious fractures in limbs
* history of metabolic or psychiatric disorder
* alcohol or drug dependency
* underlying diseases
* vegetarian diet

Ages: 16 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Glasgow Coma Scale (GCS) | 7 days
Duration of mechanical ventilation | 14 days
  Duration of mechanical ventilation is recorded by a nurse who is blinded to grouping and reported in days.
ICU stay | 14 days
Serum S100 level | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- NNFTRI clinic, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided
undecided